CLINICAL TRIAL: NCT03336398
Title: Investigation of the NMDA Antagonist Ketamine as a Treatment for Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Medical Doctor, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7432
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Ketamine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tinnitus Distressed Patients (Experimental): Tinnitus distressed patients are patients who experience symptoms of anxiety or depression with tinnitus. This group will receive both 0.5 mg/kg ketamine hydrochloride in saline and placebo, saline, with Magnetic Resonance Spectroscopy scans and audiometry testing and scales.
  Interventions: Drug: Ketamine Hydrochloride in saline; Drug: Saline
- Tinnitus Patients (Experimental): Tinnitus patients are patients who do not experience symptoms of anxiety or depression with tinnitus. This group will receive both 0.5 mg/kg ketamine hydrochloride in saline and placebo, saline, with Magnetic Resonance Spectroscopy scans and audiometry testing and scales.
  Interventions: Drug: Ketamine Hydrochloride in saline; Drug: Saline

INTERVENTIONS:
Drug: Ketamine Hydrochloride in saline — 0.5 mg/kg IV of ketamine hydrochloride in saline will be administered with one of the MRS Scan
  Other Names: Ketamine HCI
Drug: Saline — Saline will be administered with the other MRS scan
  Other Names: Saline solution

SUMMARY:
Tinnitus, or ringing in the ears, is a very common problem that often accompanies hearing loss. It affects up to 1 in 10 adults, and about 30% of people who experience chronic tinnitus find it very distressing. In these patients, symptoms of depression and anxiety often accompany tinnitus and there are no approved treatments. Clinical trials are ongoing to test a glutamate NMDA receptor antagonist (called esketamine), which is injected into the inner ear. However, the preliminary results with this medication show that it only works for tinnitus that results from acute injury. It does not treat tinnitus resulting from progressive hearing loss.

Research in humans and animals suggest that the neurotransmitters glutamate and GABA are important in the development and maintenance of tinnitus. This data shows that over-activation of the NMDA receptor and a decrease in GABA signaling in the brain play a crucial role. Previous studies show that ketamine, which an antagonist at the NMDA receptor, increases GABA levels in the brain in participants with depression. Thus, in this experiment, this study will test the effect of ketamine on tinnitus, since it blocks the NMDA glutamate receptor and increase GABA levels.

Two groups of participants will be included in this study: those who experience distress (symptoms of anxiety or depression) with tinnitus and those who have tinnitus but do not experience distress. Each participant will receive both ketamine and placebo on different days. Magnetic Resonance Spectroscopy (MRS) scans will be

DETAILED DESCRIPTION:
Tinnitus has a prevalence of approximately 1 in 10 adults in the United States. Among those with tinnitus, 36% had nearly constant symptoms and almost 30% of those report that their tinnitus as a big or a very big problem. Currently there are few effective treatments for tinnitus, and no approved medications. Cognitive behavioral and retraining therapy provide some relief, but many patients fail to respond.

Animal research and human studies indicate that maladaptive plasticity plays a role in tinnitus, which involves glutamatergic signaling largely at the NMDA and AMPA receptors. Additionally, GABA signaling has been shown to be impaired in tinnitus. Rodent models show a diminished sensitivity to GABA signaling and human magnetic resonance spectroscopy (MRS) studies show decreased GABA levels in the auditory cortex.

Ketamine is a non-competitive NMDA receptor antagonist that has also been shown to activate AMPA receptors, and modulates ongoing plasticity. Additionally, ketamine activates a subpopulation of cortical GABAergic interneurons and projection neurons and increases GABA levels in the human brain, measured with MRS. Ketamine is FDA approved as an anesthetic, and recent work has demonstrated its efficacy in treating refractory depression and chronic pain. Importantly, these demonstrate that low dose ketamine, at doses lower than those required for anesthesia, are effective in lifting depressed mood and improving the sensation of chronic pain.

For many, tinnitus has an important affective component to it, with distress and co-morbid symptoms of depression and anxiety. The onset and severity of tinnitus can correlate with stressful events, and it has been posited that stress lowers the threshold of perception, and unmasks tinnitus. Tinnitus then triggers more anxiety and depressed mood, which in turn reinforces the symptoms. An advantage of ketamine may be its effect on depression and anxiety, in addition to tinnitus, to interrupt this cycle.

The goal of this study is to perform a proof-of-concept preliminary study of ketamine in tinnitus associated with sensori-neural hearing loss. This will be studied both in participants who report depressed mood and anxiety and those who do not. MRS imaging will be used to assess ketamine-induced changes in GABA in the auditory cortex.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 21-60
* Tinnitus associated with at least mild sensori-neural hearing loss of at least 6 months duration
* Score at least 32 on the Tinnitus Handicap Inventory and a score of 5dB or greater on the minimum masking level
* Tinnitus not due to medical disease (other than sensorineural hearing loss)
* Score of at least 14 on the Hamilton Depression Rating Scales with a score of at least 2 on the Hamilton Anxiety Rating Scale (in the distressed group).

Exclusion Criteria:

* DSM-V psychiatric disorders other than mild-moderate depression and anxiety, including substance use disorder.
* History of recreational ketamine use, recreational PCP use,exposure to ketamine as an anesthetic, or an adverse reaction to ketamine
* Currently taking psychotropic medication (e.g.antipsychotics, antidepressants, benzodiazepines)
* Presence or positive history of significant medical or neurological illness, including high blood pressure (SBP >140, DBP > 90), cardiac illness, abnormality on EKG, head injury.
* Pregnancy, abortion, or lack of effective birth control during 15 days before the scan
* Metal implants, pacemaker, other metal (e.g. shrapnel or surgical prostheses) or paramagnetic objects contained within the
* Medicinal patch that cannot be removed for the scans.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in GABA and Glutamate (Glx) levels in the auditory cortex derived from 3T Magnetic Resonance Spectroscopy | during ketamine and placebo MRS scans
  The GABA and Glx peaks will be quantified as ratios

SECONDARY OUTCOMES:
Change in The Brief Psychiatric Rating Scale (BPRS) | Baseline, at the end of MRS scan, 110 minutes after ketamine or placebo infusion
  The Brief Psychiatric Rating Scale (BPRS) is a rating scale used by a clinician to measure psychiatric symptoms. The scores range from a minimum 16 to maximum of 112. Higher scores indicate a more severe disorder.
Change in The Tinnitus Handicap Inventory (THI) | screening, pre and post ketamine and placebo sessions
  The Tinnitus Handicap Inventory is a self-administered test to determine the degree of distress in tinnitus patients. Scores range from 0 to 100 with higher scores indicating a greater degree of distress from tinnitus.
Change in Visual Analogue Scale (VAS) | screening, pre and post ketamine and placebo sessions, then daily
  Visual Analogue Scale (VAS) is a scale that consists of a straight line with gradients from 0 (no tinnitus) to 10 (severe tinnitus).
  (maximal experience of tinnitus)
Change in the Beck Depression Inventory (BDI) Depression Inventory (BDI) | screening, pre and post ketamine and placebo sessions, daily for 10 days after the sessions
  The Beck Depression Inventory (BDI) is a multiple choice inventory for depression
Change in Profile of Mood States (POMS) | screening, pre and post ketamine and placebo sessions, daily for 10 days after the sessions
  The Profile of Mood States (POMS) is used to assess mood states.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Martinez, Principal Investigator — NYSPI/Columbia University
Locations (1):
- 1051 Riverside Drive, New York, New York, United States